CLINICAL TRIAL: NCT06973161
Title: External Control Arm Study for T-DXd for Patients With HER2 IHC3+ Solid Tumors (ESPERANZA)
Brief Title: ESPERANZA: External Control Arm Study for T-DXd for Patients With HER2 IHC3+ Solid Tumors
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry); Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: D967VR00001
Record Dates: First submitted 2025-04-23; First posted 2025-05-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Bladder Cancer; Biliary Tract Cancer; Cervical Cancer; Endometrial Cancer; Ovarian Cancer; Pancreatic Cancer; Colorectal Cancer; Lung Cancer; Other Tumors
MeSH Terms: conditions — Urinary Bladder Neoplasms; Biliary Tract Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Systemic Anticancer Therapy: Patients who received the existing standard of care systemic anti-cancer therapy (SACT) per routine clinical practice in the real-world setting.
- Trastuzumab Deruxtecan: Patients who received 5.4 mg/kg trastuzumab deruxtecan

SUMMARY:
In DESTINY-Pan-Tumor [DP-02], DESTINY CRC02 [DC-02], and DESTINY-Lung01 [DL-01], T-DXd demonstrated tumor response across a broad range of HER2-expressing solid tumors, particularly IHC3+ patients.

This study will use real-world data (RWD) to identify IHC3+ patients in the real world who received standard of care (SoC) and compare them with IHC3+ patients who received T-DXd in the referent trials. The tumors included are: non-small cell lung cancer [NSCLC], colorectal cancer [CRC], endometrial cancer, bladder cancer, epithelial ovarian cancer, cervical cancer, pancreatic cancer, biliary tract cancers, and other tumors.

This is a real-world external control arm (ECA) study to generate evidence on the comparative effectiveness of T-DXd versus real-world (RW) SoC in adult patients with HER2 IHC3+ solid tumors who have received prior systemic treatment. HER2 IHC3+ patients who initiated 5.4mg/kg of T-DXd in the referent trials (DP-02, DC-02, and DL-01) will be compared against IHC3+ patients who received RW SoC. This will be a retrospective observational study which will use secondary real-world data and data collected in the 3 aforementioned trials.

Objectives: The primary objective of this study is to evaluate the comparative effectiveness with respect to overall survival (OS) for T-DXd vs SoC for patients with HER2 IHC3+ expressing solid tumors in two pooled cohorts: one cohort reflecting the tumors in the three referent trials (referred to as the 'tumor agnostic' cohort), consisting of patients with NSCLC, CRC, endometrial, epithelial ovarian, cervical, pancreatic, biliary tract cancers, and other tumors; and a second cohort reflecting the tumors in the DP-02 trial (referred to as 'pan tumor'), consisting of the same tumors but excluding NSCLC and CRC.

ELIGIBILITY:
Inclusion Criteria (for the ECA):

Male or female patients aged 18 years or older at the time of locally advanced, unresectable or metastatic disease diagnosis.

Patients diagnosed with one of the following malignancies:

Locally advanced, unresectable or metastatic colorectal adenocarcinoma, biliary tract, bladder (urothelial), cervical, endometrial, epithelial ovarian, pancreatic, or other solid tumors, or unresectable and/or metastatic non-squamous NSCLC.

Patients may be included on the basis of de-novo locally advanced, unresectable or metastatic disease diagnosis or progression from initial diagnosis at earlier stages.

Patients must have received at least one line of prior systemic anti-cancer therapy (SACT) therapy in the advanced/ unresectable/ metastatic setting (i.e. excluding adjuvant/ neoadjuvant SACT) prior to index.

Index date (start of 2nd or later line SoC systemic anti-cancer therapy (SACT) treatment) for advanced disease occurring between January 2017 and December 2022.

[CRC patients only] Prior treatment at index with at least one of the following in prior lines of therapy:

Fluoropyrimidine, oxaliplatin, and irinotecan

Anti-epidermal growth factor receptor (EGFR) treatment, if RAS wild-type

Anti-vascular endothelial growth factor (VEGF) treatment

Anti-programmed death-ligand 1 (PD-[L]-1) therapy if tumor is microsatellite instable (MSI)-high/deficient mismatch repair (dMMR), or tumor mutational burden (TMB)-high

[CRC patients only] BRAF wild-type cancer and confirmed RAS status (either mutant or wild type) identified through testing of the primary tumor or metastatic site at any time following initial diagnosis.

IHC3+ HER2-expression confirmed through testing of tumor samples taken in the advanced/ recurrent/ metastatic disease stage. The sample taken closest in time prior to the or at start of the index line of therapy should be used to confirm IHC3+ HER2 status. Positive IHC3+ tests may be the result of testing at the time of sampling by the sites or retrospective testing based on archival tumor samples

ECOG of 0 or 1 (or Karnofsky score of ≥ 70%8), or missing performance status based on most recently recorded information prior to or at index date.

Patients without recorded history of liver disease, leukaemia, aplastic anaemia or haemophilia at index date.

Patients known to have died must have a complete recorded date of death.

Exclusion Criteria (for the ECA):

Record of other primary malignancies (except non-melanoma skin cancer) at any time prior to or after index.

Record of spinal cord compression prior to or at index or active CNS metastases at index (with active CNS metastases determined per physician judgment OR receipt of radiotherapy directed at CNS metastases within 6 months prior to index).

Record of myocardial infarction within 6 months prior to index date or congestive heart failure at any time prior to or at index date.

Record of lung-specific intercurrent clinically significant illness based on physician judgement prior to or at index date.

History of (non-infectious) ILD/ pneumonitis prior to or at index.

Record of autoimmune, connective tissue or inflammatory disorders prior to or at index date.

Record of complete pneumonectomy prior to or at index date.

Presence of systemic infection at index date.

Record of HIV prior to or at index date, or active Hep B or Hep C infection at index date.

Treatment with T-DXd or DXd-containing ADC at any time prior to or at index.

Record of pregnancy at or at any time following advanced/ unresectable/ metastatic disease diagnosis.

Treatment as part of a clinical trial at any time prior to or at index.

[Pan-tumor patients only] Patients with a record of pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and Concentrated Ascites Reinfusion Therapy (CART) at index.

[Colorectal patients only] Patients with record of leptomeningeal carcinomatosis prior to or at index.

[NSCLC patients only] Treatment with a HER2-targeted therapy (except for pan-HER class tyrosine kinase inhibitors) at any time prior to or at index.

[NSCLC patients only] Record of unstable angina at any time prior to or at index date.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population of interest is adult patients with HER2 IHC3+ unresectable and/or metastatic disease falling within the indications of interest. All IHC3+ patients who initiated 5.4 mg/kg of T-DXd in DP-02, DC-02, or DL-01 for each indication will be included in the T-Dxd arm of this study. To identify RW SoC patients for each indication, relevant eligibility criteria from the corresponding referent trial will be applied and modified for the RW setting where required.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Anticipated to be approximately 11 to 17 months
  Time from the date of first dose of treatment until the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (25):
- Research Site, Spartanburg, South Carolina, United States
- Research Site, Vienna, Austria
- Research Site, Liège, Belgium
- Research Site, London, Ontario, Canada
- Research Site, Olomouc, Czechia
- Research Site, Copenhagen, Denmark
- France (6):
  - Research Site, Caen
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Saint-Herblain
- Germany (4):
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Heidelberg
  - Research Site, W Rzburg
- Italy (2):
  - Research Site, Meldola
  - Research Site, Rome
- Research Site, Porto, Portugal
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Valencia
- United Kingdom (2):
  - Research Site, Leeds
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/